CLINICAL TRIAL: NCT01840020
Title: Changes in Bioavailability of Ethanol Following Bariatric Surgery
Brief Title: BAR-trial: Bioavailability of Ethanol Following Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/1206
Record Dates: First submitted 2013-04-15; First posted 2013-04-25 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Obesity, Morbid
Keywords: bariatric surgery; alcohol drinking; alcoholism; ethanol; metabolism
MeSH Terms: conditions — Obesity, Morbid; Alcohol Drinking; Alcoholism | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric bypass: patients recruited from Central Norway
  Interventions: Procedure: Gastric bypass
- Gastric sleeve: patients recruited from Central Norway
  Interventions: Procedure: gastric sleeve

INTERVENTIONS:
Procedure: Gastric bypass — Surgical procedure in which the stomach is transected high on the body. The resulting small proximal gastric pouch is joined to any parts of the small intestine by an end-to-side surgical anastomosis.
  Groups: Gastric bypass
Procedure: gastric sleeve — Sleeve gastrectomy, a surgical procedure in which the stomach is reduced to about 25% of its original size, by surgical removal of a large portion of the stomach, following the major curve. The open edges are then attached together (often with surgical staples) to form a sleeve or tube with a banana shape.
  Groups: Gastric sleeve

SUMMARY:
The first-pass metabolism (FPM) is a barrier to the toxicity of ethanol. Changes to the size and function of the stomach may alter FPM. Bariatric surgery, like the gastric bypass procedure, involves significant changes to the size and function of the stomach and leads to more rapid gastric emptying. Consequences will be faster absorption and higher peak concentration of ethanol after surgery than before. There are growing concerns that surgery for obesity in this way may cause alcohol abuse.

In this study the investigators compare changes in FPM of ethanol following two different bariatric surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* volunteers from Central Norway
* morbid obese BMI > 40 kg/m2)
* morbid obese BMI > 35 kg/m2 given a obesity related disease that qualifies for bariatric surgery

Exclusion Criteria:

* previous or current alcohol abuse
* risk for alcohol harm as assessed by AUDIT
* alcohol abstinence
* liver disease except fatty liver, which occurs in more than 50% of those who seek bariatric surgery
* previous colon resection
* not/insufficiently able to informed consent
* drugs that interact with alcohol dehydrogenase
* drugs that slow down emptying of the stomach
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: persons eligible for bariatric surgery in the Obesity policlinic, St Olavs Hospital, Trondheim, Norway
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change in bioavailability of ethanol | from baseline to 3 months, 1 year, and 3 years
  bioavailability tests: Plasma concentration of ethanol. Calculation:
  * Area under curve (AUC)
  * Maximum concentration(Cmax)
  * Time up to maximum concentration (tmax)
  * Oral bioavailability (AUCpo/AUCiv)

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Strommen, MSc, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Sykehuset Namsos, Namsos
  - Obesity policlinic of St. Olavs Hospital, Trondheim